CLINICAL TRIAL: NCT06859788
Title: Open-Label Study of SPI-1005 for the Treatment of Meniere's Disease
Brief Title: SPI-1005 for the Treatment of Meniere's Disease (Open Label)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sound Pharmaceuticals, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-1005-401
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Meniere's Disease; Ménière's Disease
Keywords: ebselen; hearing loss; tinnitus; vertigo; dizziness; SPI-1005
MeSH Terms: conditions — Meniere Disease; Hearing Loss; Tinnitus; Vertigo; Dizziness | interventions — ebselen

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): Oral administration of SPI-1005 400 mg BID
  Interventions: Drug: Ebselen

INTERVENTIONS:
Drug: Ebselen — Glutathione peroxidase mimetic
  Other Names: SPI-1005

SUMMARY:
Study of the safety of open-label SPI-1005 400 mg BID treatment in adults with Meniere's Disease (MD) for 6 or 12 months to support chronic or chronic intermittent use.

ELIGIBILITY:
Inclusion Criteria:

* Adult males/females, 18-75 years of age at the time of enrollment.
* Diagnosis of probable or definite Meniere's Disease by AAO-HNS Amended 2015 Criteria.
* At least two of three active symptoms (fluctuating hearing; tinnitus; aural fullness; vertigo or dizziness) of Meniere's disease, within 3 months of study enrollment.
* Type A tympanogram at screening.
* Air conduction thresholds ≤ 90 dB at all tested frequencies (250-8000 Hz) in both ears.
* Subject is willing and able to provide informed consent and perform study procedures and assessments per protocol.
* Reproductive requirements

Exclusion Criteria:

* Current, or within 60 days prior to study enrollment, use of IV or intratympanic ototoxic medications such as chemotherapy including cisplatin, carboplatin, or oxaliplatin; aminoglycoside antibiotics including gentamicin, amikacin, tobramycin, kanamycin, or streptomycin; or loop diuretics including furosemide.
* History of otosclerosis or vestibular schwannoma.
* History of significant middle ear or inner ear surgery in the affected ear.
* Conductive hearing loss with air-bone gap ≥15 dB, otitis media, or mixed hearing loss.
* Significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, neurological, or psychiatric disease.
* Current use or within 30 days prior to study enrollment systemic steroids.
* Current use or within 7 days prior to study enrollment intratympanic steroids.
* Hypersensitivity or idiosyncratic reaction to compounds related to ebselen or excipients.
* Female patients who are pregnant or breastfeeding.
* Participation in another investigational drug or device study within 30 days prior to study consent.
* Participant resides more than 100 miles from the study site.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 180 and 360 days
  Safety and tolerability assessed based on adverse events

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - The House Institute, Los Angeles, California
  - ENT and Allergy Associates of Florida, Boca Raton, Florida
  - University of Miami, Miami, Florida
  - Northwell Health, New Hyde Park, New York
  - ENT and Allergy Associates, LLP, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kil J, Lobarinas E, Spankovich C, Griffiths SK, Antonelli PJ, Lynch ED, Le Prell CG. Safety and efficacy of ebselen for the prevention of noise-induced hearing loss: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2017 Sep 2;390(10098):969-979. doi: 10.1016/S0140-6736(17)31791-9. Epub 2017 Jul 14. PMID 28716314
- [Background] Kil J, Pierce C, Tran H, Gu R, Lynch ED. Ebselen treatment reduces noise induced hearing loss via the mimicry and induction of glutathione peroxidase. Hear Res. 2007 Apr;226(1-2):44-51. doi: 10.1016/j.heares.2006.08.006. Epub 2006 Oct 6. PMID 17030476
- [Background] Kil J, Harruff EE, Longenecker RJ. Development of ebselen for the treatment of sensorineural hearing loss and tinnitus. Hear Res. 2022 Jan;413:108209. doi: 10.1016/j.heares.2021.108209. Epub 2021 Feb 19. PMID 33678494